CLINICAL TRIAL: NCT06017089
Title: The Pediatric Artificial Pancreas Automated Initialization Trial (PEDAP-AI): A Pilot Study of AI Advisor-Driven Pump Initiation and Parameter Adaptation in Young Children With Type 1 Diabetes
Brief Title: The Pediatric Artificial Pancreas Automated Initialization Trial
Acronym: PEDAP-AI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marc Breton (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Jaeb Center for Health Research (Other); University of Colorado, Denver (Other); Stanford University (Other)
Responsible Party: Sponsor-Investigator, Marc Breton, Principal Investigator, University of Virginia
Organization: University of Virginia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 230262; U01DK127551-03 (NIH)
Record Dates: First submitted 2023-08-18; First posted 2023-08-30 (Actual); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Continuous Glucose Monitor (CGM); Tandem t:slim Insulin Pump with Control-IQ Technology; Control-IQ Technology (CIQ); Artificial Pancreas (AP); Artificial Intelligence (AI); Closed loop control (CLC); Diabetes Assistant (DiAs)
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: In this single-arm intervention trial, all participants will use the study system (pump and CGM) in closed-loop mode for 8 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- AI Advisor-driven at-home closed loop system initiation and parameter adaptation (Experimental): In this single-arm intervention trial, all participants will use the study system (t:slim X2 with Control-IQ Technology and Dexcom Continuous Glucose Monitor) in closed-loop mode for 8 weeks at home with periodic parameter adjustment driven by an AI-based Advisor system.
  Interventions: Device: AI-based Advisor system

INTERVENTIONS:
Device: AI-based Advisor system — Tandem t:slim X2 with Control-IQ and t:connect mobile application and Dexcom G6 or G7 system, connected to UVA cloud-based Physician Dashboard with insulin pump parameters driven by an AI-based Advisor system.

SUMMARY:
The goal of this clinical trial is to obtain safety data and exploratory glycemic control data from use of an at-home closed loop control (CLC) system (t:slim X2 with Control-IQ Technology) with periodic parameter adjustments driven by an AI-based Advisor system in young children with Type 1 Diabetes. The main endpoints this study aims to answer is the safety and efficacy of the use of the AI-driven pump parameters. Participants will use the study system (pump and Continuous Glucose Monitor) in closed-loop mode for eight weeks.

DETAILED DESCRIPTION:
In this single-arm pilot study of an AI Advisor-driven closed loop system initiation and parameter adaptation in youth age 2 to <6 years old, participants will use the Tandem t:slim X2 with Control-IQ and t:connect mobile application and Dexcom G6 or G7 system, connected to the University of Virginia (UVA) cloud-based Physician Dashboard for eight weeks at home.The key safety outcomes are adverse events related to hypoglycemia and hyperglycemia, CGM-measured time spent below 54mg/dL, and CGM-measured time spent above 250 mg/dL. CGM-measured endpoints will be tested against baseline for non-inferiority.Glycemic outcomes including time in target range 70-180 mg/dL (TIR) and various other CGM measures of hypo- and hyperglycemia will be assessed and tested for superiority against baseline and a matched historical control population from the prior PEDAP study that did not involve the use of any AI-driven pump parameters. Up to 45 screened participants with the goal of at least 30 participants completing the study pump use period.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least 1 month
2. Familiarity and use of a carbohydrate ratio for meal boluses
3. Age ≥2 and <6 years old
4. Using a Dexcom CGM at the time of enrollment, with use on at least 21 out of the prior 28 days
5. Living with one or more parent/legal guardian knowledgeable about emergency procedures for severe hypoglycemia and able to contact emergency services and study staff
6. Parent/guardian has a phone that can run the Tandem t:connect Mobile App (typically Android 10 or above or iPhone Operating System (iOS) 15 or above)
7. Willingness to use the t:connect Mobile App as needed during the study and ensure connectivity for a data upload at least once per day
8. Investigator has confidence that the parent can successfully operate all study devices and is capable of adhering to the protocol
9. Willingness to switch to lispro (Humalog) or aspart (Novolog) if not using already, and to use no other insulin besides lispro (Humalog) or aspart (Novolog) during the study for participants using a study162 provided Tandem pump during the study
10. Total daily insulin dose (TDD) at least 5 Units/day
11. Body weight at least 20 pounds (lbs)
12. Willingness not to start any new non-insulin glucose-lowering agent during the course of the trial
13. Participant and parent(s)/guardian(s) willingness to participate in all training sessions as directed by study staff
14. Parent/guardian proficient in reading and writing English
15. Live in the United States, with no plans to move outside the United States during the study period

Exclusion Criteria:

1. Concurrent use of any non-insulin glucose-lowering agent (including GLP-1 agonists, Symlin, DPP-4 inhibitors, SGLT-2 inhibitors, sulfonylureas)
2. Hemophilia or any other bleeding disorder
3. History of >1 severe hypoglycemic event with seizure or loss of consciousness in the last 3 months
4. History of >1 diabetic ketoacidosis (DKA) event in the last 6 months not related to illness, infusion set failure, or initial diagnosis
5. History of chronic renal disease or currently on hemodialysis
6. History of adrenal insufficiency
7. Hypothyroidism that is not adequately treated in the opinion of the investigator
8. Use of oral or injectable steroids within the last 8 weeks
9. Known, ongoing adhesive intolerance
10. Plans to receive blood transfusions or erythropoietin injections during the course of the study
11. A condition, which in the opinion of the investigator or designee, would put the participant or study at risk
12. Participation in another pharmaceutical or device trial at the time of enrollment or during the study
13. Having immediate family members employed by Tandem Diabetes Care, Inc. or Dexcom, Inc., or having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (as a study investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the clinical trial

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Lum, MS, Study Director — Jaeb Center for Health Research; Raj P Wadwa, MD, Principal Investigator — Barbara Davis Center, University of Colorado; Marc D Breton, Ph.D., Study Chair — University of Virginia Center for Diabetes Technology
Locations (3):
- United States (3):
  - Stanford University, Stanford, California
  - Barbara Davis Center, University of Colorado, Aurora, Colorado
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Will follow the NIH Data Sharing Policy and Implementation Guidance on sharing research resources for research purposes to qualified individuals in the scientific community
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available after the primary publications of each study site.
Access Criteria: The Data Sharing Agreements will be formulated by the study team.

REFERENCES:
- [Result] Pavan J, Cobry E, Reed ZW, Villa-Tamayo MF, Diaz C JL, DeBoer MD, Schoelwer M, Jost E, Kingman R, Holmes V, Lum JW, Koravi CLK, Buckingham B, Beck R, Wadwa RP, Breton MD; PEDAP-AI Trial Study Group. Algorithm-Driven Initiation and Adaptation of Hybrid Closed-Loop in Young Children with Type 1 Diabetes: A Pilot Study. Diabetes Technol Ther. 2025 Aug;27(8):587-596. doi: 10.1089/dia.2024.0650. Epub 2025 Mar 28. PMID 40152109

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Did not meet screening eligibility (N=1)
Groups:
- AI Advisor-driven At-home Closed Loop System Initiation and Parameter Adaptation: In this single-arm intervention trial, all participants will use the study system (t:slim X2 with Control-IQ Technology and Dexcom Continuous Glucose Monitor) in closed-loop mode for 8 weeks at home with periodic parameter adjustment driven by an AI-based Advisor system.
  AI-based Advisor system: Tandem t:slim X2 with Control-IQ and t:connect mobile application and Dexcom G6 or G7 system, connected to University of Virginia (UVA) cloud-based Physician Dashboard with insulin pump parameters driven by an AI-based Advisor system.
Period: Overall Study
Arm/Group | AI Advisor-driven At-home Closed Loop System Initiation and Parameter Adaptation
Started | 32
Completed | 28
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | AI Advisor-driven At-home Closed Loop System Initiation and Parameter Adaptation
Number analyzed (Participants) | 32
Age, Customized [Count of Participants; unit: Participants]
  2 to <4 years | 9
  4 to <6 years | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 22
  More than one race | 4
  Unknown or Not Reported | 0
Body Mass Index Percentile [Median (Inter-Quartile Range); unit: percentage] | 76 [58 to 92]
Parent Education [Count of Participants; unit: Participants]
  High school graduate/diploma/GED | 4
  Technical/Vocational | 1
  Associate Degree (AA) | 4
  College Graduate (Bachelor's Degree or Equivalent) | 9
  Advanced Degree (e.g. Masters, PhD, MD) | 14
Annual Household Income [Count of Participants; unit: Participants]
  $35,000 to <$50,000 | 1
  $50,000 to <$75,000 | 5
  $75,000 to <$100,000 | 4
  $100,000 to <$200,000 | 10
  ≥$200,000 | 11
  Unknown | 1
Health Insurance [Count of Participants; unit: Participants]
  Private | 26
  Medicare | 2
  Medicaid | 4
HbA1c [Mean (Standard Deviation); unit: percentage of glycated hemoglobin] | 7.3 (0.9)
Insulin Modality [Count of Participants; unit: Participants]
  MDI | 20
  Pump | 12
Total Daily Insulin [Mean (Standard Deviation); unit: U/kg/day] | 0.61 (0.21)
Number of Pump Boluses or Injections of Short-Acting Insulin per Day [Median (Inter-Quartile Range); unit: Pump boluses per day] | 5 [3 to 6]
Diabetic Ketoacidosis (DKA) in last 12 months [Count of Participants; unit: Participants]
  No episodes | 24
  One episodes | 8
Severe hypoglycemia (SH) in Last 12 Months [Count of Participants; unit: Participants]
  None | 32
  1 | 0
Diabetes Duration [Median (Inter-Quartile Range); unit: months] | 10 [4 to 36]

OUTCOME MEASURES:

1. Primary Outcome: Safety Endpoint (Tested for Non-inferiority Compared to Baseline) CGM Measured (a)
Description: % of time below 54 mg/dL
Time Frame: Baseline and Weeks 1-8
Population: Three participants were excluded due to lack of data. To meet criteria for inclusion, participants had to provide at least 168 hours of CGM data during baseline and the 8-week follow-up period and remain in closed loop for at least 50% of the 8-week period after closed loop initiation.
Measure: Mean (Standard Deviation); unit: percentage of time
Groups:
- Baseline Period: Participants aged 2-6 years with Type 1 Diabetes were monitored using their existing insulin therapy (either multiple daily injections or personal insulin pump settings) prior to the initiation of the AI-driven intervention. Continuous glucose monitoring (CGM) data were collected for up to 28 days before the intervention to establish baseline glycemic control metrics.
- AI Advisor-driven At-home Closed Loop System Initiation and Parameter Adaptation: Participants used the Tandem t:slim X2 insulin pump with Control-IQ technology for 8 weeks. Initial and adaptive pump settings were guided by an AI-based advisor through the UVA Clinical Portal. Investigators reviewed and could override AI-generated recommendations. This period was designed to evaluate the safety and efficacy of algorithm-driven insulin delivery in a pediatric population.
Arm/Group | Baseline Period | AI Advisor-driven At-home Closed Loop System Initiation and Parameter Adaptation
Number analyzed (Participants) | 29 | 29
percentage of time | 0.3 (0.3) | 0.3 (0.2)

2. Primary Outcome: Safety Endpoint (Tested for Non-inferiority Compared to Baseline) CGM Measured (b)
Description: % of time above 250 mg/dL
Time Frame: Baseline and Weeks 1-8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Baseline Period | AI Advisor-driven At-home Closed Loop System Initiation and Parameter Adaptation
Number analyzed (Participants) | 29 | 29
percentage of time | 13 (10) | 9 (5)

3. Primary Outcome: Hierarchical Efficacy Endpoints (Tested for Superiority Compared With Baseline) CGM Measured (a)
Description: % of time in range 70-180 mg/dL
Time Frame: Baseline and Weeks 1-8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Baseline Period | AI Advisor-driven At-home Closed Loop System Initiation and Parameter Adaptation
Number analyzed (Participants) | 29 | 29
percentage of time | 63 (15) | 70 (8)

4. Primary Outcome: Hierarchical Efficacy Endpoints (Tested for Superiority Compared With Baseline) CGM Measured (b)
Description: Mean glucose
Time Frame: Baseline and Weeks 1-8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Baseline Period | AI Advisor-driven At-home Closed Loop System Initiation and Parameter Adaptation
Number analyzed (Participants) | 29 | 29
mg/dl | 168 (28) | 157 (14)

5. Primary Outcome: Hierarchical Efficacy Endpoints (Tested for Superiority Compared With Baseline) CGM Measured (c)
Description: % of time >250 mg/dL
Time Frame: Baseline and Weeks 1-8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Baseline Period | AI Advisor-driven At-home Closed Loop System Initiation and Parameter Adaptation
Number analyzed (Participants) | 29 | 29
percentage of time | 13 (10) | 9 (5)

6. Primary Outcome: Hierarchical Efficacy Endpoints (Tested for Superiority Compared With Baseline) CGM Measured (d)
Description: % of time <70 mg/dL
Time Frame: Baseline and Weeks 1-8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Baseline Period | AI Advisor-driven At-home Closed Loop System Initiation and Parameter Adaptation
Number analyzed (Participants) | 29 | 29
percentage of time | 2 (1.4) | 1.7 (0.9)

7. Primary Outcome: Hierarchical Efficacy Endpoints (Tested for Superiority Compared With Baseline) CGM Measured (e)
Description: % of time <54 mg/dL
Time Frame: Baseline and Weeks 1-8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Baseline Period | AI Advisor-driven At-home Closed Loop System Initiation and Parameter Adaptation
Number analyzed (Participants) | 29 | 29
percentage of time | 0.3 (0.3) | 0.3 (0.2)

8. Secondary Outcome: CGM Measured Time in Range
Description: % of time spent within range 70 mg/dL-140 mg/dL.
Time Frame: Baseline and Weeks 1-8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Baseline Period | AI Advisor-driven At-home Closed Loop System Initiation and Parameter Adaptation
Number analyzed (Participants) | 29 | 29
percentage of time | 42 (14) | 47 (9)

9. Secondary Outcome: CGM Measured (a)
Description: % of time >180 mg/dL
Time Frame: Baseline and Weeks 1-8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Baseline Period | AI Advisor-driven At-home Closed Loop System Initiation and Parameter Adaptation
Number analyzed (Participants) | 29 | 29
percentage of time | 35 (15) | 29 (8)

10. Secondary Outcome: CGM Measured (b)
Description: % of time >300 mg/dL
Time Frame: Baseline and Weeks 1-8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Baseline Period | AI Advisor-driven At-home Closed Loop System Initiation and Parameter Adaptation
Number analyzed (Participants) | 29 | 29
percentage of time | 5.9 (5.6) | 3.3 (2.6)

11. Secondary Outcome: CGM Measured (c)
Description: % of time <60 mg/dL
Time Frame: Baseline and Weeks 1-8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Baseline Period | AI Advisor-driven At-home Closed Loop System Initiation and Parameter Adaptation
Number analyzed (Participants) | 29 | 29
percentage of time | 0.7 (0.5) | 0.6 (0.4)

12. Secondary Outcome: CGM Measured (d)
Description: Glucose standard deviation
Time Frame: Baseline and Weeks 1-8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Baseline Period | AI Advisor-driven At-home Closed Loop System Initiation and Parameter Adaptation
Number analyzed (Participants) | 29 | 29
mg/dl | 64 (16) | 59 (12)

13. Secondary Outcome: CGM Measured (e)
Description: Glucose coefficient of variation
Time Frame: Baseline and Weeks 1-8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Baseline Period | AI Advisor-driven At-home Closed Loop System Initiation and Parameter Adaptation
Number analyzed (Participants) | 29 | 29
percent | 38 (5) | 37 (5)

14. Secondary Outcome: CGM Measured (f)
Description: The high blood glucose index (HBGI) is based on a nonlinear transformation of blood glucose values that corrects for the asymmetry of the glucose scale. This transformation maps glucose values into a risk space (minimum risk = 0), where higher values correspond to higher risk. Values below 10 suggest low to moderate risk.
Time Frame: Baseline and Weeks 1-8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Baseline Period | AI Advisor-driven At-home Closed Loop System Initiation and Parameter Adaptation
Number analyzed (Participants) | 29 | 29
index | 8.8 (5) | 6.8 (2.5)

15. Secondary Outcome: CGM Measured (g)
Description: The low blood glucose index (LBGI) is based on a nonlinear transformation of blood glucose values that corrects for the asymmetry of the glucose scale. This transformation maps glucose values into a risk space (minimum risk = 0), where higher values correspond to higher risk. Values <1 suggest low risk of hypoglycemia.
Time Frame: Baseline and Weeks 1-8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Baseline Period | AI Advisor-driven At-home Closed Loop System Initiation and Parameter Adaptation
Number analyzed (Participants) | 29 | 29
index | 0.6 (0.4) | 0.6 (0.2)

16. Secondary Outcome: CGM Measured (h)
Description: Weekly hyperglycemic event rate
Time Frame: Baseline and Weeks 1-8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Baseline Period | AI Advisor-driven At-home Closed Loop System Initiation and Parameter Adaptation
Number analyzed (Participants) | 29 | 29
events | 1.9 (2.0) | 1.1 (1.0)

17. Secondary Outcome: CGM Measured (i)
Description: Weekly hypoglycemic event rate
Time Frame: Baseline and Weeks 1-8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Baseline Period | AI Advisor-driven At-home Closed Loop System Initiation and Parameter Adaptation
Number analyzed (Participants) | 29 | 29
events | 0.6 (0.6) | 0.4 (0.4)

18. Secondary Outcome: Binary Outcome 1
Description: Number of participants whose % of time in range 70-180 mg/dL improved by 5% or more from baseline to 8 weeks.
Time Frame: Baseline and Weeks 1-8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- AI Advisor-driven At-home Closed Loop System Improvement From Baseline: Participants used the Tandem t:slim X2 insulin pump with Control-IQ technology for 8 weeks. Initial and adaptive pump settings were guided by an AI-based advisor through the UVA Clinical Portal. Investigators reviewed and could override AI-generated recommendations. This period was designed to evaluate the safety and efficacy of algorithm-driven insulin delivery in a pediatric population.
Arm/Group | AI Advisor-driven At-home Closed Loop System Improvement From Baseline
Number analyzed (Participants) | 29
Participants | 13

19. Secondary Outcome: Binary Outcome 2
Description: Number of participants whose % of time in range 70-180 mg/dL improved by 10% or more from baseline to 8 weeks.
Time Frame: Baseline and Weeks 1-8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AI Advisor-driven At-home Closed Loop System Improvement From Baseline
Number analyzed (Participants) | 29
Participants | 9

20. Secondary Outcome: Binary Outcome 3
Description: Participants with % of time in range 70-180 mg/dL >70% and % of time <70 mg/dL <4%
Time Frame: Baseline and Weeks 1-8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline Period | AI Advisor-driven At-home Closed Loop System Initiation and Parameter Adaptation
Number analyzed (Participants) | 29 | 29
Participants | 10 | 13

21. Secondary Outcome: Total Daily Insulin
Description: Total daily insulin (units/kg)
Time Frame: Baseline and Weeks 1-8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/kg
Arm/Group | Baseline Period | AI Advisor-driven At-home Closed Loop System Initiation and Parameter Adaptation
Number analyzed (Participants) | 29 | 27
U/kg | 0.59 (0.20) | 0.66 (0.19)

22. Secondary Outcome: Basal Insulin
Description: Percentage of total insulin delivered via basal administration.
Time Frame: Baseline and Weeks 1-8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of total insulin
Arm/Group | Baseline Period | AI Advisor-driven At-home Closed Loop System Initiation and Parameter Adaptation
Number analyzed (Participants) | 29 | 27
percentage of total insulin | 39 (17) | 38 (9)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | AI Advisor-driven At-home Closed Loop System Initiation and Parameter Adaptation
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 3/32
Other Adverse Events (participants affected / at risk) | 5/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AI Advisor-driven At-home Closed Loop System Initiation and Parameter Adaptation (N=32)
Severe Hypoglycemia (Endocrine disorders) | 1 (1) — severe hypoglycemic event is defined as a hypoglycemic event that a) required assistance of another person due to altered consciousness, and b) required another person to actively administer carbohydrate, glucagon, or other resuscitative actions
Diabetic Ketoacidosis (Endocrine disorders) | 1 (1) — Hyperglycemia: Blood glucose level ≥ 250 mg/dL (13.9 mmol/L) Ketosis: Presence of moderate to large ketonuria or Serum β-hydroxybutyrate ≥ 3.0 mmol/L Metabolic Acidosis: Arterial or venous pH < 7.3 and/or Serum bicarbonate < 15-18 mmol/L
Other serious adverse events (Endocrine disorders) | 1 (1) — Hypoglycemia due to user error when changing infusion set.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AI Advisor-driven At-home Closed Loop System Initiation and Parameter Adaptation (N=32)
Hyperglycemia with or without Ketosis (Endocrine disorders) | 3 (3)
Gastroenteritis (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/89/NCT06017089/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT06017089/SAP_001.pdf
  • Informed Consent Form (2024-03-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT06017089/ICF_002.pdf